CLINICAL TRIAL: NCT07236268
Title: Prevalence of HIV and Sexually Transmitted Infections in Migrant Communities in Slovakia With a Special Emphasis on Refugees From Ukraine
Brief Title: Prevalence of HIV and Sexually Transmitted Infections in Migrant Communities in Slovakia
Status: Completed | Type: Observational
Sponsor: Comenius University (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Alexandra Brazinova, Chair of Institute of Epidemiology, Faculty of Medicine, Comenius University
Other Study IDs: 2023/1338156-0
Record Dates: First submitted 2025-11-15; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: STIs; HIV; Rapid Detection
Keywords: STI rapid screening; HIV screening; Hepatitis C screening; Syphilis screening; Hepatitis B screening
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 - volunteers at outpatient healthcare facility: Patients coming to visit general practitioner or gynaecologist (at outpatient healthcare facility serving Ukrainian war refugees residing temporarily in Bratislava region) who underwent voluntary free-of-charge screening for HIV, syphilis, hepatitis B and C by rapid test based on a capillary blood drop from a fingerpick.
- Group 2 - volunteers at health screening event: Persons participating at community health screening one day event for Ukrainian war refugees residing temporarily in Bratislava region.

SUMMARY:
Before project launch, key materials were prepared, including informed consents, posters, informational leaflets, patient cards, social media posts, standard operating procedures, patient management plans and patient registries. Necessary medical supplies (rapid tests for HIV, syphilis, hepatitis B and C, lancets, sterile pads, gloves and personal protective equipment) were secured.

The main field activity took place at the Health Care Centre for Ukrainian refugees in Bratislava (Rovniankova 1), operated by EQUITA and the Bratislava Administrative Region. The screening offer was promoted through posters, leaflets distributed to patients, and social media channels (Facebook, Instagram, Telegram). Testing was provided during regular operating hours to all patients.

A psychologist was available throughout the project to support patients with reactive results, help arrange appointments for laboratory confirmation and specialist care, and accompany patients if requested. Confirmatory diagnostics and treatment pathways were pre-arranged with University Hospital Bratislava (Dermatovenerology Clinic for syphilis; Infectious Diseases Clinic for HIV and viral hepatitis).

Rapid testing using capillary blood was conducted. Participants signed informed consent before testing. Four drops of finger-prick blood were applied to rapid test plates, with results available after 10 minutes. Patient IDs, anonymized codes and results were recorded. Regardless of results, all patients received basic counselling on the screened diseases and prevention. In reactive cases, patients were informed immediately, referred for confirmation, and provided psychological support. Confirmed patients received clinical evaluation and treatment covered by state health insurance. Medical and administrative supplies at the facility were replenished weekly.

A second field activity, "Health Day," was implemented at the Assistance Centre on Bottova Street, operated by the Municipality of Bratislava. Partners included the Regional Public Health Authority, the Bratislava Association of Medical Students and SCORA, and EQUITA. The event was promoted through posters and social media. Participants were offered rapid testing for HIV, syphilis, hepatitis B and C, as well as basic cardiovascular screening and stool tests for occult bleeding. Informational brochures, condoms, menstrual aids and patient cards were distributed.

DETAILED DESCRIPTION:
Before launching the project, all required materials were prepared, including informed consents, posters, informational leaflets, patient cards, social media posts, standard operating procedures, patient management plans and registries. Medical supplies (rapid tests for HIV, syphilis, hepatitis B and C, lancets, sterile pads, gloves and PPE) were secured.

The main field activity took place at the Health Care Centre for Ukrainian refugees in Bratislava (Rovniankova 1), operated by EQUITA and the Bratislava Administrative Region. Screening was promoted through posters in waiting areas, printed leaflets, and social media (Facebook, Instagram, Telegram). Testing was provided during regular operating hours to any patient. A psychologist was present to support reactive cases and assist with referral and follow-up. Prior agreements ensured laboratory confirmation and specialist care at University Hospital Bratislava (Dermatovenerology for syphilis; Infectious Diseases Clinic for HIV, hepatitis B and C).

Rapid screening using capillary finger-prick blood was conducted. After informed consent, four blood drops were applied to rapid tests, with results available in 10 minutes. Patient identifiers, anonymized codes and results were recorded. All patients received basic prevention counselling. Reactive patients were immediately informed, referred for confirmatory testing, and guided to specialist care; therapy was covered by state health insurance. Supplies at the Centre were replenished weekly.

A second field activity, "Health Day," was implemented at the Assistance Centre on Bottova Street in cooperation with multiple partners. The event offered rapid testing for HIV, syphilis, hepatitis B and C, basic cardiovascular screening, and colorectal cancer stool tests. Informational materials, condoms and menstrual aids were distributed, and participants received patient cards documenting results.

ELIGIBILITY:
Inclusion Criteria:

* Ukrainian war refugees residing temporarily in Bratislava region, 18 years and older, signing the informed consent

Exclusion Criteria:

* non Ukrainian war refugees, age less than 18 years, not signing the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ukrainian war refugees residing temporarily in Bratislava region, 18 years and older, that after signing the informed consent underwent rapid screening test for HIV, syphilis, hepatitis B and C. All participants with reactive results were offered consultation with a psychologist and were referred to specialist for laboratory diagnosis and treatment.
Sampling Method: Non-Probability Sample
Enrollment: 660 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
HIV, syphilis, hepatitis B, hepatitis C reactivity rates | From enrolment to 9 months after enrolment
  Reactive result on rapid screening

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Bražinová, prof. MD, PhD, Principal Investigator — Comenius University, Faculty of Medicine, Institute of Epidemiology
Locations (1):
- Comenius University, Faculty of Medicine in Bratislava, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No